CLINICAL TRIAL: NCT05568771
Title: The Effect of The Modified Injury Prevention Program Asisted With Core Strength Training on Anaerobic Power And Core Strength in Young Women Basketball Players
Brief Title: Core Strength Training on Anaerobic Power And Core Strength in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Core Strenght and Anaerobic
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core exercise group (Experimental): In the study, the exercise group was set as Istanbul University Club Basketball Team, and the control group was set as Galatasaray Basketball Club. While the 1st group, which is the exercise group, applied the additional warm-up program to the core training program to be included in the routine training of the team, for 8 weeks,
  Interventions: Other: Core Exercises Assisted Injury Prevention Training Program
- Control group (No Intervention): the 2nd group, the control group, continued their routine training programs.

INTERVENTIONS:
Other: Core Exercises Assisted Injury Prevention Training Program — After the exercises are fully taught to the athletes, the core training program will be applied on 3 non-consecutive days of the week, accompanied by a physiotherapist or athletic trainer, and the warm-up program will be applied before all trainings of the team, except before the match.The core program will take 20-25 minutes, and the warm-up program will take an average of 20-25 minutes. The exercises consist of an average of 45 minutes. This warm-up program includes running exercises, strengthening exercises, balance and proprioception exercises, and plyometric exercises.
  Arms: Core exercise group

SUMMARY:
The aim of the study is to investigate the effect of injury prevention program with core strength training support on anaerobic power and core strength in woman basketball Players In this direction, it is expected that the program will contribute to the decrease in the incidence of injury, the vertical jump distance, which is an indicator of anaerobic power, and the increase of core muscle strength.

DETAILED DESCRIPTION:
This study was approved by the ethics committee of Istanbul University Istanbul Faculty of Medicine.It will be done in the Exercise Test Laboratory of the Department of Medicine.

Istanbul University youth women's basketball team and Galatasaray youth women's youth basketball teams will be included in the study.The Vertical Jump test, Cybex Isokinetic Core Strength Assessment will be measured before and after the 8-week exercise training for both the study and control group.The sample group of the study was found to be 40 people as a result of the statistical analysis made with reference to the peak torque.

First of all, people will be informed about the "Informed Voluntary Consent Form" and the study will be explained. Then, volunteers who agree to participate in the study and meet the criteria for participation in the study will be asked to read the "Informed Voluntary Consent Form" or sign it themselves or their legal guardians.

Athletes will be distributed into two groups by randomization method. The 1st group (working group) will apply the additional warm-up program to the core training program, which will be included in the routine training of the team, for 8 weeks, the 2nd group (control group) will continue their routine training programs.

Cybex Isokinetic Core Force Assessment: Core strength will be evaluated using Cybex HUMAC/NORM (CSMI, 2004) brand isokinetic equipment, which measures torque produced against different speeds. With the isokinetic machine, the body extension-flexion movement will be measured with an angle of 60° and 90°. Similar to athletic performance tests, subjects will also complete a practice session on the machine prior to the test. Prior to core strength tests, subjects will warm up on the treadmill at low speeds for approximately 10 minutes for warm-up purposes. Trunk extension-flexion and measurements will be obtained following Smith et al.'s procedures.Verbal support will be provided by subjects to encourage maximum effort. Any report of symptoms of pain, shortness of breath, and/or dizziness will be recorded during the testing session.

The range of motion will be adjusted from 10° extension to 45° flexion (ROM: 55°).

Mutually concentric trunk flexion and extension will be evaluated at 60°/sec and 90°/sec angular velocities.

During each trial, five repetitions of submaximal warm-ups will be performed before each test rate. A 5-second rest period will be allowed between the warm-up reps and the actual test session. For the test procedure, five maximum concentric contractions will be performed at an angular rate of 60°/sec. To test durability, 15 repetitions will be used at an angular rate of 90°/sec. The tests will begin in the full extension position. There will be a 20 second rest period between each angular speed test.

They will be verbally encouraged during the test session to show maximum physical effort.

* Peak torque (Newton-meter (Nm)): It is the highest force value produced by the muscle. It can be determined at each repetition during the movement. Peak torque can be evaluated according to a certain time or angle (EHA) throughout the movement. Since peak torque is an absolute value, it may be insufficient in the evaluation alone and the same values may be interpreted differently from person to person.
* The ratio of peak torque to body weight (Newton.Meter/Kilogram): It is the ratio of the maximum torque produced to body weight. The heavier of two people with equal peak torque value will have a lower Peak torque/body weight ratio, while the one with the lower weight will have a higher value. This value will be evaluated according to sport activity, function, age and gender.
* Time to reach peak torque (seconds): It is the time for the muscle to reach maximum force. It indicates the ability of the muscles to produce maximum torque quickly.
* Peak torque reaching angle (degrees): It is the point where the peak torque is produced at the angle scanned throughout the movement.

Vertical Jump Test: University of Toronto Belt Jump (Sports Books Publisher, Toronto, Ontario, Canada) consists of a rubber mat on which the participant stands and a tape feeder in the middle. The tape measure will be attached to a belt that is tied around the participant's waist. The bottom of the tape measure will pass through a feeder combined with the mat and the tape measure will be adjusted 0 cm before the jump. The tape measure will slide along the feeder until the participant reaches the top of the jump. After the jump, the height from the length of the tape pulled from the feeder will be recorded.

They will perform a total of six jumps, with a maximum of three for warm-up before data collection. Specifically, subjects will do 2 sets of 10 repetitions each of the "arm swing", "lunge walking", "'walking knee lift" and "heel to toe lift" warm-ups before the test.

Before each jump, participants will be instructed to "stand upright" for 3 seconds on the corresponding measuring device, which includes standing completely upright with their shoulders back and arms at their sides to standardize the starting position. At the end of this period, participants will be reminded to jump to the maximum level before being instructed to "jump". At the end of this period, participants will be reminded to jump to the maximum level before being instructed to "jump". They will then perform a maximum counter-motion jump (CMJ) with arm swing. If a participant jumps forward from the landing area, the jump will be repeated.

Exercise Training After the exercises are fully taught to the athletes, the core training program will be applied on 3 non-consecutive days of the week, accompanied by a physiotherapist or athletic trainer, and the warm-up program will be applied before all trainings of the team, except before the match. In the 1st group training program, progress will be made in the exercises in the 2,5, v 8th weeks. The exercises selected for the core exercise program will be performed by creating stations from easy to difficult, with the help of the "Developing the core" book. As for the warm-up program, a combined protocol was created by considering the FIFA+11 and FIFA+11 S programs. The core program will take 20-25 minutes, and the warm-up program will take an average of 20-25 minutes. The exercises consist of an average of 45 minutes. This warm-up program includes running exercises, strengthening exercises, balance and proprioception exercises, and plyometric exercises.

In the shoulder External Rotation/Internal Rotation strengthening exercises that will be applied between 0-2 weeks, the arms will be adjacent to the trunk.2-5. arm 45 degrees in weeks, 5-8. In weeks, the arm is abducted 90 degrees. Low weights will be preferred in the exercises, and while the upper extremity exercises are planned to be performed 3 sets of 10-15 repetitions, the progress will be made by increasing the resistance and weights. Lower extremity exercises including exercises such as running, balance and proprioception will be performed 2 times for 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 15-24
* Being cooperative,

Exclusion Criteria:

* The athlete has a history of diagnosed orthopedic, neurological or musculoskeletal disease that interferes with assessments,
* Having undergone a surgical operation in the last 6 months,
* There is a situation that prevents you from training.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Anaerobic Power | 15 minute
  Maximal power (work per unit time) developed during all-out, short-term physical effort; reflects energy-output capacity of intramuscular high-energy phosphates (ATP and PCr) and/or anaerobic glycolysis, Anaerobic power was evaluated with the vertical jump test.
Core Strength | 20 minute
  the strength of the underlying muscles of the torso, which help determine posture. The strength of the core muscles was evaluated with an isokinetic device.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent BAYRAKTAR, Prof, Principal Investigator — Istanbul University; Ömer Bayrak, Study Director — Istanbul University
Locations (1):
- Istanbul University Sport Medicine Department, Fatih, Turkey (Türkiye)

REFERENCES:
- [Result] Karatas GK, Gogus F, Meray J. Reliability of isokinetic trunk muscle strength measurement. Am J Phys Med Rehabil. 2002 Feb;81(2):79-85. doi: 10.1097/00002060-200202000-00001. PMID 11807340
- [Result] Buckthorpe M, Morris J, Folland JP. Validity of vertical jump measurement devices. J Sports Sci. 2012;30(1):63-9. doi: 10.1080/02640414.2011.624539. Epub 2011 Nov 23. PMID 22111944
- [Result] Baechle, T.; Earle, R.W.; Wathen, D. Resistance Training. In Essentials of Strength Training and Conditioning; Baechle, T., Earle, R., Eds.; Human Kinetics: Champaign, IL, USA, 2008